CLINICAL TRIAL: NCT04221074
Title: Ultrasound Guided Modified Pectoral Plane (PECS II )Block Versus Erector Spinae Plane (ESP) Block for Perioperative Analgesia of Surgical Treatment of Gynecomastia
Brief Title: Ultrasound Guided Modified Pectoral Plane Block Versus Erector Spinae Plane Block During GA in Gynecomastia Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, manal mohamed rashad, lecturer of anaesthesia, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N B in gynecomastia surgery
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Gynecomastia, Adolescent
MeSH Terms: conditions — Gynecomastia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Pectoral Plane (PECSII ) block (P) (Active Comparator): done after induction of general anaesthesia in supine position of the patient with his arm of the side of the operation abducted 90 degree with the probe with frequency L4-12t (Logiq e machine) at the midclavicular level and angled infero-laterally,the axillary artery and vein and the second rib identified the probe moved laterally until the pectoralis minor and serratus anterior are identified,the local anesthetic was injected at two points using (echoplext guge20 length 50 mm ) needle:the first injection of 10 ml of 0.25% Bupivacaine and 4 mg dexamethasone injected between the pectoralis major and minor muscles,and the second injection of 20 ml of 0.25% Bupivacaine and 4 mg dexamethasone between the pectoralis minor and serratus anterior muscles .
  Interventions: Procedure: PECS II versus ESP
- Erector Spinae Plane ( ESP )block (E) (Active Comparator): after induction of general anaesthesia in lateral position of the patient where the surgical side up and at T4 level the probe with frequency L4-12t (Logiq e machine) placed lateral to the spine by 3 cm in parasagittal plane the needle (echoplext guge20 length 50 mm ) advanced between the transverse process and the erector spinae muscle at that level 20 ml of 0.25% Bupivacaine and 8 mg dexamethasone injected.
  Interventions: Procedure: PECS II versus ESP

INTERVENTIONS:
Procedure: PECS II versus ESP — compare between :ultrasound guided Pectoralis nerve(pecs) II block or erector spinae plane (ESP) block in surgical treatment for gynecomastia patients under general anaesthesia.

SUMMARY:
Pain of breast surgery is due to chest wall scar and arm in some cases like carcinoma or due to nerve injury.It is neuropathic or nociceptive pain.Its severity is depending on the extent of surgery and the radiotherapy if needed.

Previous studies proved that local nerve block procedures improved the immediate postoperative pain and decreased the incidence of postoperative pain chronicity .

Also effective control of pain suppresses the surgical stress response minimizes the anaesthestic needs intraoperatively and decreases the opioid needs postoperatively .

Pectoralis nerve(pecs) II block and erector spinae plane (ESP) block are novel procedures that may provide good intraoperative and postoperative analgesia in patients undergoing surgical treatment of gynecomastia.

ELIGIBILITY:
Inclusion Criteria:

* Male gender .
* Age : 18 - 25 years old .
* Physical status : ASA I - II .
* Body mass index(BMI) :20-30 kg/m2
* Surgical treatment of Gynecomastia .
* Duration of surgery : 60 -120 min

Exclusion Criteria:

* Patient refusal .
* History of opioid abuse or chronic analgesic use .
* Coagulopathy .
* Allergy to study drugs .
* Infection in the injection sites.
* Uncooperative patients.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
intraoperative analgesia | 60-120 minuets
  measurement of intraoperative mean blood pressure (mmHg)
intraoperative analgesia | 60-120 minuets
  measurement of heart rate (beat /min)
intraoperative analgesia | 60-120 minuets
  measurement of bispectral index score

SECONDARY OUTCOMES:
postoperative analgesia | 24 hours
  evaluation of postoperative visual analogue scaleusing a ruler graded from 0 to 100 mm,where 0=no pain and 100=the worst imaginable pain measured in postanaesthesia care unit and every 6hours for 24 h postoperative.
postoperative analgesia | 24 hours
  time interval till first analgesic request (minuets)
postoperative analgesia | 24 hours
  total opioid consumption (mg)

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university, Zagazig, Egypt